CLINICAL TRIAL: NCT01457846
Title: A Randomised Open-Label Phase II Study to Assess the Efficacy & Safety of AZD4547 Monotherapy Versus Paclitaxel in Patients With Advanced Gastric Adenocarcinoma (Inc. Adenocarcinoma of the Lower Third of the Oesophagus or the Gastro-Oesophageal Junction)With FGFR2 Polysomy or Gene Amplification.
Brief Title: Efficacy and Safety of AZD4547 Versus Paclitaxel in Patients With Advanced Gastric or Gastro-oesophageal Cancer
Acronym: SHINE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D2610C00004
Record Dates: First submitted 2011-09-16; First posted 2011-10-24 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Gastro-oesophageal Junction Cancer; Gastric Cancer
Keywords: gastro-oesophageal junction cancer; gastric cancer; lower third oesophageal cancer; polysomy; amplification; FGFR
MeSH Terms: conditions — Stomach Neoplasms | interventions — AZD4547; Paclitaxel

ARMS (2):
- AZD4547 (Experimental): AZD4547 taken orally in tablet formation, 80mg b.d., in a 2 week on, 1 week off schedule
  Interventions: Drug: AZD4547
- Paclitaxel (Active Comparator): Paclitaxel - 80mg/m² as a 1 hour infusion given weekly on days 1, 8 and 15 of a 28 day cycle (up to the maximum number of cycles per local practice)
  Interventions: Drug: paclitaxel

INTERVENTIONS:
Drug: AZD4547 — Tablets taken, oral, twice daily, commencing with a 2 week on AZD4547, 1 week off AZD4547 schedule.
  Arms: AZD4547
Drug: paclitaxel — Infusion administered once a week, 3 weeks on and 1 week off
  Arms: Paclitaxel

SUMMARY:
The purpose of this study is to assess the efficacy, safety and tolerability of AZD4547 compared with paclitaxel in patients with advanced gastric or lower-oesophageal cancer whose tumours are found to have FGFR2 polysomy or gene amplification.

DETAILED DESCRIPTION:
A Randomised Open-Label Phase IIa Study to Assess the Efficacy and Safety of AZD4547 monotherapy versus paclitaxel in Patients with Advanced Gastric or Gastro-oesophageal Junction Cancer with FGFR2 Polysomy or Gene Amplification (SHINE study). Patients were to be assigned to strata by FGFR2 status of: polysomy, low or high gene amplification.

ELIGIBILITY:
Inclusion Criteria:

* Female or male aged 25 or over
* Histological diagnosis of locally advanced or metastatic gastro adenocarcinoma (including adenocarcinoma of the lower third of the oesophagus or the gastro oesophageal junction )
* Radiographically confirmed progression after 1 prior chemotherapy or chemoradiotherapy for gastric cancer. Suitable for and expected to benefit from paclitaxel monotherapy.
* At least one lesion, not previously irradiated, that has baseline at least 10mm in the longest diameter for non nodal lesions and is assessed by Computerised Tomography (CT) or Magnetic Resonance Imaging (MRI)
* Provision of either an archival tumour sample or a fresh tumour sample for confirmation of FGFR2 polysomy/gene amplification

Exclusion Criteria:

* Prior exposure to AZD4547 or history of hypersensitivity other drugs similar in structure or class to AZD4547. Hypersensitivity to paclitaxel or formulated in cremophor EL (polyoxyethylated castor oil)
* Prior taxane treatment for gastric cancer with the exception of adjuvant/neo-adjuvant therapy given > 6 months; Major surgery, radiotherapy with wide field of radiation or any cancer treatment within 4 weeks before the first dose of the study treatment
* With the exception of alopecia, any unresolved toxicities from prior therapy with a Common Terminology Criteria for AE (CTCAE) grade >1 at the time of starting study treatment.
* Blood and Echocardiogram (ECG) readings that are deemed to be abnormal by falling outside of the reference ranges in the protocol inclusion/exclusion section.
* Taking other regular medication that are predicted to interact with AZD4547 due to their route of metabolism.

Ages: 25 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 960 (Actual)
Dates: Start 2011-11; Primary Completion 2013-08 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Stockman, MD PHD, Study Director — AstraZeneca; Eric Van Cutsem, MD PHD, Principal Investigator — University Hospital, Gasthuisberg; Yung-Jue Bang, MD, PHD, Principal Investigator — Seoul National University Hospital
Locations (61):
- Belgium (4):
  - Research Site, Brussels (Anderlecht)
  - Research Site, Brussels (Woluwé-St-Lambert)
  - Research Site, Leuven
  - Research Site, Liège
- Bulgaria (3):
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Vratsa
- Canada (2):
  - Research Site, Fredericton, New Brunswick
  - Research Site, Toronto, Ontario
- Czechia (3):
  - Research Site, Brno
  - Research Site, Olomouc
  - Research Site, Prague
- France (2):
  - Research Site, Saint-Cloud
  - Research Site, Villejuif
- Germany (2):
  - Research Site, Hamburg
  - Research Site, Mainz
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Nyíregyháza
- India (6):
  - Research Site, Bangalore
  - Research Site, Chennai
  - Research Site, Hyderabad
  - Research Site, Nagpur
  - Research Site, Pune
  - Research Site, Vellore
- Italy (4):
  - Research Site, Ancona
  - Research Site, Milan
  - Research Site, Pisa
  - Research Site, Roma
- Japan (6):
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Kōtoku
  - Research Site, Nagoya
  - Research Site, Sapporo
  - Research Site, Takatsuki-shi
- Romania (2):
  - Research Site, Brasov
  - Research Site, Cluj-Napoca
- South Korea (6):
  - Research Site, Anyang-si
  - Research Site, Daegu
  - Research Site, Hwasun-gun
  - Research Site, Jeonju
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (6):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Oviedo
  - Research Site, Santander
  - Research Site, Seville
- Taiwan (4):
  - Research Site, Keelung
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Ukraine (2):
  - Research Site, Kharkiv
  - Research Site, Lviv
- United Kingdom (6):
  - Research Site, Aberdeen
  - Research Site, London
  - Research Site, Maidstone
  - Research Site, Manchester
  - Research Site, Sutton
  - Research Site, Wolverhampton

REFERENCES:
- See also: D2610C00004redacted_protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1284&filename=D2610C00004_ProtocolCSP_2Redactions_marked14Dec15_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 11 countries. Enrolment started in November 2011 and last patient visit was in August 2013. In total, 960 patients were enrolled out of which 71 were randomised. A total of 67 patients received treatment , 40 of these patients received AZD4547 and 27 received Paclitaxel.
Pre-assignment Details: Patients ≥ 25 years with locally advanced or metastatic gastric adenocarcinoma that had FGFR2 polysomy or FGFR2 gene amplification and whose disease had progressed during or after 1st line therapy. Patients whose disease had progressed within 6 months following adjuvant or neo-adjuvant therapy could be included at the discretion of the investigator
Groups:
- AZD4547: 80mg BD 2 weeks on/1 week off
- Paclitaxel: 80mg / m^2
Period: Overall Study
Arm/Group | AZD4547 | Paclitaxel
Started | 41 | 30
Received Treatment | 40 | 27
Did Not Receive Treatment | 1 | 3
Ongoing Treatment at Data Cut-off | 1 | 1
Completed | 0 | 0
Not Completed | 41 | 30
Not completed — Death before treatment | 1 | 2
Not completed — Did not receive treatment | 0 | 1
Not completed — Death | 27 | 16
Not completed — Unclassified reason for not completed | 11 | 10
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paclitaxel | AZD4547 | Total
Number analyzed (Participants) | 30 | 41 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at time of screening
  years | 61.9 (10.65) | 60.6 (11.38) | 61.2 (11.02)
Age, Customized [Number; unit: Participants]
  <50 years | 4 | 7 | 11
  >=50 - < 65 years | 13 | 20 | 33
  >= 65 years | 13 | 14 | 27
Gender [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 22 | 29 | 51

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival
Description: PFS is the time from randomisation until the date of objective disease progression as defined by Response Evaluation Criteria In Solid Tumours (RECIST version 1.1) or death (by any cause in the absence of progression).
Time Frame: Tumour size assessed at week 8 (±1 week) and then every 8 weeks (±1 week)
Population: Full analysis set
Measure: Number; unit: months
Arm/Group | AZD4547 | Paclitaxel
Number analyzed (Participants) | 41 | 30
months | 1.8 | 3.5
Statistical Analysis 1: Comparison: AZD4547 vs Paclitaxel; Test type: Superiority or Other; p = 0.9581, Regression, Cox — 1-sided; Hazard Ratio (HR) = 1.57, 80% CI 2-sided [1.12 to 2.21]

2. Secondary Outcome: Overall Survival : Number of Patients Who Had Died at DCO (Data Cut Off)
Time Frame: Tumour size assessed at week 8 (±1 week) and then every 8 weeks (±1 week)
Population: This secondary analysis included factors for treatment and FGFR2 FISH score (4/5 versus 6) and is based on the Full analysis set (all treated patients).
Measure: Number; unit: Patients
Arm/Group | AZD4547 | Paclitaxel
Number analyzed (Participants) | 38 | 30
Patients | 27 | 18
Statistical Analysis 1: Comparison: AZD4547 vs Paclitaxel; Test type: Superiority or Other; p = 0.8156, Regression, Cox — 1-sided; Hazard Ratio (HR) = 1.31, 80% CI 2-sided [0.89 to 1.95]

3. Secondary Outcome: Objective Response Rate
Description: ORR=Percentage of patients with at least one visit response of CR (complete response) or PR (partial response) that is confirmed at least 4 weeks later; CR:disappearance of target lesions and no new lesions; PR is at least 30% decrease in sum of diameters of lesions taking as a reference the smallest sum since treatment started.
Time Frame: Week 8 (±1 week) and then every 8 weeks (±1 week)
Population: The analysis included factors for treatment and FGFR2 FISH score (4/5 versus 6) and is based on the Full analysis set (all treated patients).
Measure: Number; unit: Patients (%)
Arm/Group | AZD4547 | Paclitaxel
Number analyzed (Participants) | 38 | 30
Patients (%) | 2.6 | 23.3
Statistical Analysis 1: Comparison: AZD4547 vs Paclitaxel; Test type: Superiority or Other; p = 0.9970, Regression, Logistic — 1-sided; Odds Ratio (OR) = 0.09, 80% CI 2-sided [0.02 to 0.35]

4. Secondary Outcome: Percentage Change From Baseline at Week 8 in Target Lesion Size
Description: A negative change denotes a reduction in target lesion size. Percentage change from baseline in tumour size at 8 weeks in target lesion size.
Time Frame: Baseline, Week 8 (±1 week)
Population: Full analysis set - all treated patients with at least one post baseline RECIST target lesion assessment scan
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | AZD4547 | Paclitaxel
Number analyzed (Participants) | 36 | 26
Percentage change | 28.4 (44.4) | -1.1 (36.18)

5. Secondary Outcome: Percentage of Patients Without Progressive Disease at 8 Weeks
Description: PD = A ≥ 20% increase in the sum of diameters of target lesions and an absolute increase of ≥ 5mm, taking as reference the smallest sum of diameters since treatment started including the baseline sum of diamters
Time Frame: Week 8 (±1 week)
Population: Full analysis set - all treated patients
Measure: Number; unit: Percentage of patients
Arm/Group | AZD4547 | Paclitaxel
Number analyzed (Participants) | 41 | 30
Percentage of patients | 24.4 | 53.3

ADVERSE EVENTS:
Time Frame: AEs will be collected throughout the study, from randomisation until the end of the follow-up period. The follow-up period is defined as 28 days after study treatment (AZD4547 or paclitaxel) is discontinued.
Arm/Group | AZD4547 | Paclitaxel
Serious Adverse Events (participants affected / at risk) | 8/40 | 6/27
Other Adverse Events (participants affected / at risk) | 39/40 | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD4547 (N=40) | Paclitaxel (N=27)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arterial disorder (Vascular disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Transaminases increases (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD4547 (N=40) | Paclitaxel (N=27)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 6 (6)
Detatchment of retinal pigment epithelium (Eye disorders) | 6 (6) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (10) | 6 (6)
Fatigue (General disorders) | 6 (6) | 8 (8)
Diarrhoea (Hepatobiliary disorders) | 6 (6) | 6 (6)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
Aspartate aminotransferase (Investigations) | 7 (7) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 16 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 13 (13)
Urinary tract infections (Infections and infestations) | 2 (2) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 9 (9)
Dry eye (Eye disorders) | 4 (4) | 0 (0)
Macular degeneration (Eye disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (8) | 5 (5)
Oedema peripheral (General disorders) | 4 (4) | 2 (2)
Asthenia (General disorders) | 11 (11) | 5 (5)
Stomatis (Gastrointestinal disorders) | 10 (10) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 9 (9) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 1 (1)
Blood phosphorus increased (Investigations) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)
Lethargy (Nervous system disorders) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 6 (6) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Onychomadesis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Onycholysis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 10 (10) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 9 (9) | 5 (5)
Dry mouth (Metabolism and nutrition disorders) | 9 (9) | 0 (0)
Alanine aminotransferase increased (Investigations) | 6 (6) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 2 (2)
Neuropathy peripheral (Psychiatric disorders) | 1 (1) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
Prompted by slow recruitment, AZ and the SRC instigated unscheduled analysis of the efficacy and tolerability. It was concluded that the study was unlikely to meet its primary objective. Enrolment ceased and the study closed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less